CLINICAL TRIAL: NCT05561647
Title: Quantitative Testing of Patient and Prescriber Knowledge About GATTEX (Teduglutide) for Injection Safety and Use Information
Brief Title: A Survey to Assess Participants' and Physicians' Knowledge When Using GATTEX (Knowledge Assessment Survey)
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-633-4008; EUPAS48716 (Registry Identifier: EU PAS Registry)
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Short Bowel Syndrome (SBS)
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GATTEX: Participants: Participants who have taken GATTEX in the 60 days prior to survey implementation are eligible to participate in this Risk Evaluation and Mitigation Strategy (REMS) survey via internet, telephone, and paper.
  Interventions: Other: No Intervention
- GATTEX: Healthcare Providers (Prescribers): HCPs (adult and pediatric) in the United States (US) who have prescribed GATTEX at least once regardless of their completion of the voluntary GATTEX REMS training are eligible for participation in this REMS survey via internet, telephone, and paper.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is non-interventional study.

SUMMARY:
The study is about learning and documenting how well participants and physicians understand how to use GATTEX and about potential risks by using a survey (called Knowledge Assessment Survey). This survey, which is conducted every two years, is part of the Gattex Risk Evaluation and Mitigation Strategy (REMS). REMS is a safety program required by the US health authority (FDA) for certain medicines that have serious risks. REMS intends to help reduce these risks while still allowing treatment. The goal is to make sure these medicines are used in the safest way possible. The main aim of this survey is to find out how well participants and physicians understand the checkups and tests (so called monitoring) participants should have while taking GATTEX, and the possible risks or of using GATTEX to treat Short Bowel Syndrome.

The knowledge assessment survey will be done via internet, telephone, or paper and both physicians and participants will be able to choose the method that is preferred.

No study medicines will be provided to participants in this study.

ELIGIBILITY:
Participant inclusion criteria:

Participants who are 18 years of age and who have taken GATTEX in the 60 days prior to survey implementation are eligible to participate in the survey. A caregiver may participate in this survey on behalf of a participant who is eligible but unable to complete the survey. Note: Participants who have previously participated in a GATTEX Patient Knowledge Assessment Survey, are eligible.

Prescriber inclusion criteria:

HCPs (adult and pediatric) in the United States who can provide a 10-digit National Provider Identifier (NPI) number and who have prescribed GATTEX at least once regardless of their completion of the voluntary GATTEX REMS training (Prescriber Education Slide Deck) are eligible for participation in the survey. Note: HCPs who have previously participated in a GATTEX Prescriber Knowledge Assessment Survey, are eligible

Participant and Prescriber exclusion criteria:

* Respondents who do not agree to participate in the survey.
* Respondents who are currently working for and/or whose immediate family members who are currently working for Takeda Pharmaceuticals U.S.A., Inc., NPS Pharmaceuticals, Inc., Shire, UBC, or the Food and Drug Administration (FDA) are not eligible to participate in the survey.
* Respondents who reported having a conflict of interest.
* HCPs who have opted out of receiving communications about the GATTEX Prescriber Knowledge Assessment Survey for the current wave

Further details associated with respondents who do not meet the exclusion criteria established above, will be provided in the assessment report.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants and prescriber who have completed Wave 8 of the GATTEX Knowledge Assessment Survey will be observed in this REMS survey.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-08-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants and Prescribers Providing Correct Responses to Questions | Up to 18 years
  All questions for survey knowledge domain and about GATTEX will be asked through a questionnaire, Participant or HCPs would need to respond true or false to each question based upon understanding and knowledge. Respondents could be participants or HCPs.

SECONDARY OUTCOMES:
Number of Participants and Prescribers Providing At Least 80 Percent (%) Correct Responses to Each Survey Knowledge Domains | Up to 18 years
  The questions will be asked to participants and HCPs and will be counted as correct if 80% of the correct responses are provided and not more than 1 incorrect response is provided. In each survey knowledge domain, general questions about GATTEX will be asked; participants or HCPs would need to respond true or false to each question based upon understanding and knowledge. Respondents could be participants or HCPs.
Number of Participants and Prescribers who Demonstrated Understanding of Survey Knowledge Domains | Up to 18years
  Understanding demonstration is defined as respondents who answered 80% or more questions/items in a survey knowledge domain correctly. In each survey knowledge domain, general questions about GATTEX will be asked, and participants or HCPs would need to respond true or false to each question based upon understanding and knowledge. Respondents could be participants or HCPs.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Pharmaceuticals, U.S.A., Inc., Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/43674fa3720540ed?idFilter=%5B%22TAK-633-4008%22%5D